CLINICAL TRIAL: NCT06038773
Title: Social and Clinical Aspects of Pelvic Pain in Turkey
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: Yeditepeu3
Record Dates: First submitted 2023-09-07; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Chronic Pelvic Pain Syndrome
MeSH Terms: interventions — Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnosis — Baseline data were presented with descriptive statistics. Sociodemographic information, pregnancy status, surgical history, exercise habits, gynecologic, obstetric, urologic and gastrointestinal history of the patients were evaluated with the "Patient Information Form".Pain intensity was evaluated with the McGill pain questionnaire short form. At the same time, the patients drew the areas where they felt the most pain with the pain maps scale. Pain intensity during sexual intercourse was evaluated with the Visual Analog Scale (VAS).Sexual Abuse Items on the Questionnaire (Modified from Badgley).

SUMMARY:
Chronic Pelvic Pain (CPP) is a common medical condition with a complex treatment due to different variables that influence its clinical course.There is a growing literature which discussing the effect of ethnicity and culture on pain. It was aimed to invesitigate whether there is a considerable difference in the presentation and experience of pelvic pain in women from a different societies and cultures.

DETAILED DESCRIPTION:
Chronic Pelvic Pain (CPP) is a common medical condition with a complex treatment due to different variables that influence its clinical course.There is a growing literature which discussing the effect of ethnicity and culture on pain. It was aimed to invesitigate whether there is a considerable difference in the presentation and experience of pelvic pain in women from a different societies and cultures.

The study includes randomly selected 45 females who completed a comprehensive set of questions derived from International Pelvic Pain Society (IPPS), pelvic pain assesment form. Character and intensity of pain, sexual abuse and harresment, coping with pain, physical activites (exercising) and comorbidities were evaluated. The McGill pain questionnaire short form was used to evaluate pain. Sexual Abuse Items in the Questionnaire (modified) to assess patients' sexual abuse status.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-65 years with pelvic pain ≥6 months were eligible.

Exclusion Criteria:

* Patient who have had pelvic surgery
* Gynecological female patients with problems other than pelvic pain

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included 45 women with pelvic pain. Women aged 18-65 years with pelvic pain ≥6 months were eligible. The study was conducted at Yeditepe University Hospital on female patients diagnosed with chronic pelvic pain syndrome due to pelvic floor muscle problems by a gynecologist.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
McGill pain scale | 1 month
  ".Pain intensity was evaluated with the McGill pain questionnaire short form. At the same time, the patients drew the areas where they felt the most pain with the pain maps scale.

CONTACTS AND LOCATIONS:
Overall Officials: nilüfer cerbezer, Msc, Principal Investigator — Yeditepe Üniversitesi
Locations (1):
- Nilüfer Cerbezer, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided